CLINICAL TRIAL: NCT04702204
Title: Efficacy and Safety of Denosumab Treatment in Bisphosphonate Unresponsive Postmenopausal Osteoporotic
Brief Title: Efficacy of Denosumab Treatment in Bisphosphonate Unresponsive Patients
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Ercan KAYDOK, Asst. Prof. MD., Nigde Omer Halisdemir University
Other Study IDs: 123
Record Dates: First submitted 2021-01-03; First posted 2021-01-08 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Denosumab 60 MG/ML — Denosumab, another antiresorptive agent, is a fully human monoclonal IgG2 antibody that binds to the receptor activator of the nuclear factor-kB ligand (RANKL) with high specificity and affinity. Denosumab inhibits bone resorption by affecting the development, activation, and survival of osteoclasts.
  Denosumab 60 mg subcutaneously was administered to the patients whose consent forms were obtained, once every 6 months.

SUMMARY:
This study, which was designed as a prospective observational study, was planned to enroll 75 female patients with postmenopausal osteoporosis who had been using bisphosphonates for more than two years and did not respond to treatment. 2 doses of denosumab were administered to the patients every 6 months. Bone mineral density of patients were measured with DEXA at the beginning and end of the study. A total of 66 patients completed the study.

At the end of the study, there was a significant improvement in the femur and lumbar total bone mineral density of the patients compared to the baseline. However, no statistically significant difference was found in terms of the frequency of new fractures.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman with postmenopausal osteoporosis
* Being between the ages of 45-85
* Using bisphosphonate therapy for at least two years
* Vertebral and/or Femur T score below -2.5
* Unresponsive to bisphosphonate therapy

  * More than 2% decrease in BMD values despite using bisphosphonates and/or
  * New major fracture development during treatment

Exclusion Criteria:

* Male gender
* Being extremely thin (BMI <15) or extremely obese (BMI> 45)
* Malignancy
* Severe chronic liver and kidney failure
* Chronic Steroid use
* Having an active rheumatic disease
* Having other secondary causes of osteoporosis (primary hyperparathyroidism etc.).

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because denosumab treatment only has FDA approval for postmenopausal osteoporosis.
Study Population: This study, which was designed as a prospective observational study, was planned to enroll 75 female patients with postmenopausal osteoporosis who had been using bisphosphonates for more than two years and did not respond to treatment.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 12 month
  Femur and spine bone mineral density measurements of the patients at the baseline and the 12th month were performed using the Dual Energy X-ray Absorptiometry (DEXA) machine (Stratos dR 2D Fan-Beam, DMS company, France).

SECONDARY OUTCOMES:
Major Bone Fracture | 12 month
  number of newly developed vertebral and femur fractures during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Bor FTR Education and Training hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 13. Miller PD, Pannacciulli N, Malouf-Sierra J, Singer A, Czerwiński E, Bone HG, et al. Efficacy and safety of denosumab vs. bisphosphonates in postmenopausal women previously treated with oral bisphosphonates. Osteoporos Int. 2020;31(1):181-91. 14. Kamimura M, Nakamura Y, Ikegami S, Uchiyama S, Kato H, Taguchi A. Significant improvement of bone mineral density and bone turnover markers by denosumab therapy in bisphosphonate-unresponsive patients. Osteoporos Int. 2017;28(2):559-66. 15. Roux C, Hofbauer LC, Ho PR, Wark JD, Zillikens MC, Fahrleitner-Pammer A, et al. Denosumab compared with risedronate in postmenopausal women suboptimally adherent to alendronate therapy: efficacy and safety results from a randomized open-label study. Bone. 2014;58:48-54 16. von Keyserlingk C, Hopkins R, Anastasilakis A, Toulis K, Goeree R, Tarride JE, et al. Clinical efficacy and safety of denosumab in postmenopausal women with low bone mineral density and osteoporosis: a meta-analysis. Semin Arthritis Rheum. 2011;41(2):178-86.